CLINICAL TRIAL: NCT04158180
Title: Creation and Validation of a Questionnaire on Diastasis Recti Signs and Symptoms
Brief Title: Creation and Validation of a Questionnaire Evaluating Diastasis Recti
Acronym: QUEDIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: QUEDIA
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2022-11

CONDITIONS: Diastasis Recti and Weakness of the Linea Alba; Diastasis Recti
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questionnaire — A battery of questionnaires will be propose to the participants

SUMMARY:
Introduction. Distasis rectus abdominis (DRA) is defined as the presence of divergence between the rectus abdominis muscles along the linea alba. Some authors describe a prevalence of 40% in women up to one year postpartum. Some studies suggest that the presence of DRA can be related to the appearance of low back, pelvic and abdominal pain and even urinary incontinence. These factors can significantly affect the quality of life of women with diastasis both socially, sexual and personal level. According to several studies, this pathology is related to higher rates of depression and an alteration in the self-perception of body image that makes these women to look to specialized medical care.

At present, the quantitative evaluation of DRA is performed purely anatomically. This evaluation consists in measuring the separation between the two rectus abdominis. Currently there is no consensus as to the protocol that should be used for this measurement.

So far, no instrument is able to quantitatively measure the consequences of DRA. The evaluation of symptoms and consequences should include relevant parameters such as quality of life, perception of body image and functional limitations.

The objective of this study is the creation and validation of a specific questionnaire to evaluate the symptoms and consequences of DRA.

Material and methods. A) Development of the questionnaire

1. Literature review
2. Online survey
3. Expert panel
4. Pilot test of the questionnaire

B) Validation of the questionnaire. The psychometric properties of the questionnaire will be evaluated in a sample of patients with DRA. The sample will be composed of a group of adult women with DRA who attended to a physiotherapy clinic.

DETAILED DESCRIPTION:
Introduction. Women with Diastasis rectus abdominis (DRA) often experience decreased physical health and functioning, negative body image and abdominal discomfort. These parameters have major impact on quality of life, becoming an additional barrier to physical activity during pregnancy and postnatal period. Nowadays, the most utilized method to evaluate DRA consists of measuring the separation between the two medial borders of the rectus abdominis muscles (namely inter-recti distance). Nevertheless, any specific tool has been created for the evaluation of parameters such as quality of life, body image perception, pain and secondary functional limitations. A valid and reliable instrument, with acceptable psychometric properties is necessary to specifically evaluate symptoms of DRA and to improve the evaluation of DRA and ultimately improve patient-centered care.

The main aim of this projet is the development and validation of such a tool.

Material and methods.

The current project consists of several stages:

A) Development of the questionnaire.

1. Literature review. A systematic review will be created to identify the relevant self-reported variables in the study of DRA in adult women. Observational studies evaluating the link between DRA and self-reported symptoms will be searched through Medline, Embase, and Cochrane Library databases. The methodological quality will be assessed independently by two evaluators using the NIH Quality Assessment Tool for Observational Cohort and Cross-Sectional Studies. This review was registered in Prospero (Review Registration Number: PROSPERO CRD42017058089). This systematic review will be conducted in accordance with the PRISMA statement.
2. Online survey. A mixed observational study will be performed through a semi-structured online survey in order to identify relevant variables in women with DRA. The Ethics Committee of the University of Valencia (June 5, 2019, 13.49.17) approved the implementation of this study. Women will sign an informed consent. The study will be carried out in accordance with the Declaration of Helsinki. The analysis of the perception of the symptoms of DRA and its repercussion at a physical, psychological and social level in women affected by this condition will be assessed. The data will be analyzed quantitatively and qualitative. Key concepts will be categorized according to their dimension through the International Classification of Functioning, Disability and Health (ICF).The CHERRIES publication guideline will be used to report the survey data.
3. Expert panel. Taking in account the results of both, the systematic review and the online survey, a first generation of items will be performed by the main authors. These items will be presented in a panel composed by various experts in this field (with prominent academic background or an extended work experience related with DRA management and/or research methods) and a patient. Experts will rate the comprehensiveness, relevance, and coherence of each item in a 4-points numerical scale. They will categorized each item in the dimension to which they believed it appertained. Aiken´s V index will be calculated. A preliminary version of the Questionnaire will be then created.
4. Pilot test of the questionnaire. The preliminary version of the Questionnaire will be tested in a pilot sample composed of 30 females with DRA. The Ethics Committee of the University of Valencia (June 5, 2019, 13.49.17) and the Committee at Canterbury Christ Church University (10/08/2021 ETH2021-0362) approved the implementation of this study. Women will sign an informed consent. The study will be carried out in accordance with the Declaration of Helsinki. Women will complete a set of questions including demographic data, the preliminary questionnaire and an evaluation of the preliminary questionnaire. An evaluation of the comprehensibility, comprehensiveness and relevance of each item will be performed using a 4-point Likert scale. Participants will be able to include their comments and remarks, individually for each item, as well as for the whole questionnaire and the questionnaire structure. Final version of the questionnaire will be then created. After the completion of the study, the dataset will be published. The COSMIN Study Design checklist for Patient-reported outcome measurement instruments will be used to report and design this study.

B) Validation of the questionnaire. The psychometric properties of the questionnaire will be evaluated in a sample of patients with DRA. The sample will be composed of a group of adult women with DRA who attended to a physiotherapy clinic. Participants will complete a series of questions including sociodemographic variables and the final version of the questionnaire. In order to calculate convergent validity, participants will be asked to complete five comparative questionnaires: Whoqol-bref overall quality of life and general health" subscale, GIQLI "Symptoms" subscale, Whoqol-bref "social relationships" subscale, WHODAS-36 "mobility" and "life activities" subscales and Body Image States Scale (BISS).Internal consistency, the type error, the ceiling floor effect, the convergent validity, the validity of the construct, the discriminatory capacity and the minimum detectable change of the questionnaire will be calculated. Seven to 10 days after the completion of the online survey, participants will be asked to fill in the final questionnaire again in order to evaluate test-retest reliability. The standard error of the measurement, the minimum detectable change and the intraclass correlation coefficient will be calculated. After the completion of the study, the dataset will be published. The COSMIN Study Design checklist for Patient-reported outcome measurement instruments will be used to report and design this study.

ELIGIBILITY:
Inclusion Criteria:

* subjects with diastasis recti,
* adult,
* women.

Exclusion Criteria:

* cognitive disabilities that can difficult a good understanding of the questionnaire,
* lack of knowledge of Spanish language.
* ventral hernia.
* previous abdominal surgeries.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult women with diastasis recti attending to a physiotherapist or midwive center will be proposed to participate in the study. A signed informed consent will be necessary to participate in this research.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Diastasis abdominal consequences | 7 to 10 days after initial assessment
  Diastasis rectus abdominis consequences will be measured using the Diastasis rectus abdominis questionnaire

SECONDARY OUTCOMES:
Inter-recti distance | Initial assessment
  The distance between the two medial borders of rectus abdominis muscles will be measured using ultrasound
Subjective well-being | Initial assessment
  Subjective well-being will be measured using the World Health Organization Quality-of-Life Scale (WHOQOL-Bref) "overall quality of life and general health" subscale (2-10 points). Domain scores are scaled in a positive direction, higher scores denote higher quality of life.
Gastrointestinal symptoms | Initial assessment
  Gastrointestinal symptoms will be measured using the Gastrointestinal Quality of Life Index (GIQLI) "Symptoms" subscale (0-36 points). 4-likert scale ( 0 points being the worst punctuation and 4 points the best)
Functioning | Initial assessment
  Functioning will be measured using the World Health Organization Disability Assessment Schedule-36 (WHODAS-36) "mobility" and "life activities"subscales (0-36points). 5- point Likert scale. Higher scores indicate lower quality of life.
Body image | Initial assessment
  Body image will be measured using the Body Image States Scale (BISS) (6-54points). The scale was presented in a negative-to-positive direction for half of the items and a positive-to-negative direction for the other half.
Social relationships-related quality of life | Initial assessment
  Social relationships-related quality of life will be measured using the World Health Organization Quality-of-Life Scale (WHOQOL-bref) "social relationships" subscale (3-15 points). Domain scores are scaled in a positive direction, higher scores denote higher quality of life.
Psychological distress | Initial assessment
  Psychological distress will be measured using Kessler psychological distress scale (K10). Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress. (10-50 points)

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Rejano Campo, PhD(c), Principal Investigator
Locations (2):
- Spain (2):
  - Haro&Campos Physiotherapy., Plasencia, Cáceres
  - Department of Physiotherapy. University of Valencia, Valencia